CLINICAL TRIAL: NCT00278525
Title: Trial of High Dose Cyclophosphamide and Rabbit Antithymocyte Globulin (rATG) With Hematopoietic Stem Cell Support in Patients With Systemic Scleroderma: A Randomized Trial
Brief Title: Cyclophosphamide and rATG With Hematopoietic Stem Cell Support in Systemic Scleroderma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Richard Burt, MD, MD, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DI Scl.Randomized2004
Record Dates: First submitted 2006-01-15; First posted 2006-01-18 (Estimated); Results first posted 2014-04-30 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-03

CONDITIONS: SYSTEMIC SCLERODERMA
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Standard of Care; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- stem cell trasplantation (Experimental): intervention as stem cell transplantation after conditioning regimen
  Interventions: Procedure: stem cell transplantation
- standard of care (Active Comparator): medication as standard of care will be given
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: standard of care — standard of care medication will be given
  Arms: standard of care
Procedure: stem cell transplantation — The following is intervention: stem cell transplantation after conditioning regimen
  Other Names: stem cell transplant, stem cell injection
  Arms: stem cell trasplantation

SUMMARY:
Scleroderma is a systemic disorder categorized as an immunologically mediated disease that causes collagen deposition of skin and visceral organs. The molecular pathogenesis of scleroderma has been elusive, although vasculopathy and immune mediated mechanisms are thought to be important. Once extensive cutaneous or visceral disease occurs, prognosis is significantly shorter than the general population. Although various treatments have been tried, none of them seems to have changed the natural history of scleroderma. Standard dose immunosuppressive treatment has been disappointing. Recently, cyclophosphamide at 1-2 mg/kg/day orally or 800-1400 mg intravenous (IV) monthly for 6-9 months has proven effective in treatment of scleroderma alveolitis (1). Recent phase I studies of immunoablation with autologous peripheral blood stem cell transplantation (PBSCT) showed some promising data, but the exact efficacy is undetermined (2,3). We now propose, as a phase II randomized study, autologous unmanipulated PBSCT versus pulse cyclophosphamide in patients with systemic scleroderma.

DETAILED DESCRIPTION:
To evaluate the efficacy of two treatment modalities: pulse cyclophosphamide versus high dose cyclophosphamide and anti-thymocyte globulin (ATG) rescued with autologous peripheral blood stem cell transplantation (PBSCT). The primary endpoints to be considered in this study are:

I)Time to Treatment Failure -Treatment failure will not occur until a minimum of 12 months after enrollment at which time failure is defined as:

1. Failure of skin score (if > 14 on enrollment) to improve or increase in skin score by a 25% above lowest post treatment value and must be documented on 2 occasion 6 months apart
2. Deterioration in diffusing capacity of the lung for carbon monoxide (DLCO), diffusing capacity divided by the alveolar volume (DLCO/VA) or forced vital capacity (FVC) by 10% below enrollment level or 10% below best post treatment value, due to systemic sclerosis, and documented on 2 occasion 6 months apart
3. Renal failure due to systemic sclerosis and defined as chronic dialysis for more than 12 months
4. Gastrointestinal failure due to systemic sclerosis and defined as initiation of total parenteral nutrition (TPN) for more than 12 months

II) Disease improvement defined by at least 25% improvement in skin score (Rodnan), or 10% improvement in pulmonary function tests (DLCO, DLCO/VA, or FVC), or in cardiac tests [pulmonary artery (PA) systolic pressure by right heart cath) that persists > 6 months or ability to wean off TPN

ELIGIBILITY:
Inclusion Criteria:

* Age 60 year or < 60 year old at the time of pretransplant evaluation.
* An established diagnosis of scleroderma.
* Diffuse cutaneous scleroderma with involvement proximal to the elbow or knee and a Rodnan score of > 14

AND

Scleroderma with any one of the following:

* Diffusing capacity of the lung for carbon monoxide (DLCO) < 80% of predicted or decrease in lung function [DLCO, diffusing capacity divided by the alveolar volume (DLCO/VA) or forced vital capacity (FVC) ] of 10% or more over 12 months.
* Active alveolitis on bronchoalveolar lavage.
* Pulmonary fibrosis or alveolitis on computed tomography (CT) scan or chest x-ray (CXR) (ground glass appearance of alveolitis).
* Renal disease that is not explained by a bacterial infection or other renal disorders. (Subjects must have two or more of the following: proteinuria - greater than trace on dipstick, hematuria - urine blood on dipstick or sediment, hypertension that requires treatment with anti-hypertensive medications or untreated but with a diastolic blood pressure (BP) > 95 mm/hg.)
* Abnormal electrocardiogram (EKG) (non-specific ST-T wave abnormalities, low QRS voltage, or ventricular hypertrophy), or pericardial effusion or pericardial enhancement on magnetic resonance imaging (MRI)
* Gastrointestinal tract involvement confirmed on radiological study. Radiologic findings of scleroderma are small bowel radiographs showing thickened folds with dilated loops, segmentation, and flocculation +/- diverticulae, or pseudodiverticulae. A hide-bound appearance due to valvulae packing i.e. dilated and crowded circular folds, may be present. Gastrointestinal (GI) involvement may also be confirmed by D-xylose malabsorption, patulous esophagus, or esophageal manometry.

OR

As published in NEJM, 2006, 345:25 2655-2709. Limited or diffuse SSL with lung involvement defined as active alveolitis on bronchoalveolar lavage (BAL) or ground-glass opacity on CT, a DLCO < 80% predicted or decrease in lung function (DLCO/VA,DLCO, FVC) of 10% or more in last 12 months.

Exclusion Criteria:

* Poor performance status Eastern Cooperative Oncology Group (ECOG 2) at the time of entry.
* Significant end organ damage such as:

  1. Left Ventricular Ejection Fraction (LVEF) < 40% or deterioration of LVEF during exercise test on Multiple Gated Acquisition (MUGA) or echocardiogram.
  2. Untreated life-threatening arrhythmia.
  3. Active ischemic heart disease or heart failure.
  4. End-stage lung disease characterized by total lung capacity (TLC) <45% of predicted value.
  5. Pulmonary hypertension (systolic pulmonary arterial pressure > 40 mmHg or mean pulmonary arterial pressure (PAP) > 25 mmHG measurement by pulmonary arterial catheter).
  6. Serum creatinine > 2.0 mg/dl.
  7. Liver cirrhosis, transaminases > 3x of normal limits or bilirubin > 2.0 unless due to Gilberts disease.
  8. Pericardial effusion> 200ml unless successful pericardiocentesis
  9. Tricuspid annular peak systolic excursion (TAPSE) ≤ 1.9 cm
  10. MRI of heart showing D sign (intraventricular flattering)
* Human immunodeficiency virus (HIV) positive.
* Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive treatment.
* Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as (but not limited to) head and neck cancer, or stage I or II breast cancer will be considered on an individual basis.
* Positive pregnancy test, inability or unable to pursue effective means of birth control, failure to willingly accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* Inability to give informed consent.
* Major hematological abnormalities such as platelet count < 100,000/ul or absolute neutrophil count (ANC) < 1000/ul.
* Patients with duration of disease > 5 years.
* Exclude if > than 6 prior monthly IV cyclophosphamide treatments.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2005-09; Primary Completion 2011-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Feinberg School of Medicine, Chicago, Illinois, United States

REFERENCES:
- [Derived] Bruera S, Sidanmat H, Molony DA, Mayes MD, Suarez-Almazor ME, Krause K, Lopez-Olivo MA. Stem cell transplantation for systemic sclerosis. Cochrane Database Syst Rev. 2022 Jul 29;7(7):CD011819. doi: 10.1002/14651858.CD011819.pub2. PMID 35904231
- [Derived] Burt RK, Shah SJ, Dill K, Grant T, Gheorghiade M, Schroeder J, Craig R, Hirano I, Marshall K, Ruderman E, Jovanovic B, Milanetti F, Jain S, Boyce K, Morgan A, Carr J, Barr W. Autologous non-myeloablative haemopoietic stem-cell transplantation compared with pulse cyclophosphamide once per month for systemic sclerosis (ASSIST): an open-label, randomised phase 2 trial. Lancet. 2011 Aug 6;378(9790):498-506. doi: 10.1016/S0140-6736(11)60982-3. Epub 2011 Jul 21. PMID 21777972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible (n=19) Randomized (n=19)
  1. Allocated to Hematopoietic Stem Cell Transplantation (HSCT (n=10) + crossed over to HSCT(n=7)
     • Received HSCT (n=17); Lost to follow-up (n=0); Analysed (n=17)
  2. Allocated to cyclophosphamide (n=9) • Received allocated intervention (n=9) Lost to follow-up (n=0); Crossed over (n=7); Analysed (n=9)
Groups:
- Standard of Care: Cyclophosphamide will be given as approved immunosuppressive therapy
Period: Overall Study
Arm/Group | Standard of Care | Stem Cell Trasplantation
Started | 9 | 10
Completed | 9 (7 participants crossed to HSCT arm in accordance with the protocol) | 10 (7 participant crossed over to the HSCT arm and underwent HSCT, in accordance with the protocol.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stem Cell Trasplantation | Standard of Care | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 9 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (13) | 44 (10) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure
Description: -Data are reporting number of participants that were classified as treatment failures
  Time to Treatment Failure Definition-Treatment failure will not occur until a minimum of 12 months after enrollment at which time failure is defined as:
  1. Failure of skin score (if > 14 on enrollment) to improve or increase in skin score by a 25% above lowest post treatment value and must be documented on 2 occasion 6 months apart
  2. Deterioration in diffusing capacity of the lung for carbon monoxide (DLCO), diffusing capacity divided by the alveolar volume (DLCO/VA) or forced vital capacity (FVC) by 10% below enrollment level or 10% below best post treatment value, due to systemic sclerosis, and documented on 2 occasion 6 months apart
  3. Renal failure due to systemic sclerosis and defined as chronic dialysis for more than 12 months
  4. Gastrointestinal failure due to systemic sclerosis and defined as initiation of total parenteral nutrition(TPN) for more than 12 months
Time Frame: 12 months
Population: All participants were included
Measure: Number; unit: participants
Groups:
- Standard of Care: Intravenous (IV) will be given 1000 mg/m2 cyclophosphamide monthly for 6 months.
Arm/Group | Stem Cell Trasplantation | Standard of Care
Number analyzed (Participants) | 10 | 9
participants | 0 (0.01) | 8 (0.11)

2. Primary Outcome: Disease Improvement
Description: Data are reporting number of participants that were classified as disease improvement.
  Definition of disease improvement:
  Disease improvement defined by at least 25% improvement in skin score (Rodnan), or 10% improvement in pulmonary function tests [diffusing capacity of the lung for carbon monoxide (DLCO), diffusing capacity divided by the alveolar volume (DLCO/VA), or forced vital capacity (FVC)], or in cardiac tests [pulmonary artery (PA) systolic pressure by right heart cath] that persists > 6 months or ability to wean off total parenteral nutrition (TPN)
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Stem Cell Trasplantation | Standard of Care
Number analyzed (Participants) | 10 | 9
participants | 10 | 0

ADVERSE EVENTS:
Time Frame: 100 days after the transplant
Description: Common Toxicity Criteria Scale used to grade all non-hematologic toxicities
Arm/Group | Stem Cell Trasplantation | Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/9
Other Adverse Events (participants affected / at risk) | 7/17 | 3/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Trasplantation (N=17) | Standard of Care (N=9)
Positive stool culture for Clostridium difficile (Infections and infestations) | 1 (1) | 0 (0) — During hospitalisation for transplantation, 1 patient had a positive stool culture for Clostridium difficile
Positive blood culture for micrococcus (Infections and infestations) | 1 (1) | 0 (0) — During the hospitalisation for transplantation, 1 patient had a positive blood culture for micrococcus
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) — During hospitalisation for transplantation, one patient developed Supraventricular tachycardia that was controlled with oral medication
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) — During hospitalisation for transplantation, 1 patient developed Atrial fibrillation that was controlled with oral medication
Volume overload (Cardiac disorders) | 2 (2) | 0 (0) — During the hospitalization for transplantation, two patients developed volume overload that were controlled with diuretics
Cytomegalovirus reactivation on surveillance blood test (Infections and infestations) | 1 (1) | 0 (0) — The only one infectious event after hospitalisation for transplantation was a cytomegalovirus reactivation on surveillance blood test in one patent, which was treated with oral valganciclovir.
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) — One patient in the control group developed cellulitis that was treated with oral antibiotics.
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 2 (2) — Two patients from the control group needed protracted outpatient treatment for gastroenteritis with nausea, vomiting and diarrhoea

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes